CLINICAL TRIAL: NCT00360958
Title: Ultrafiltration for the Chronic Treatment of Severe Congestive Heart Failure
Brief Title: Treatment of Severe Heart Failure by Ultrafiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, MD PhD, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCM S67/306
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Severe Congestive Heart Failure
Keywords: ultrafiltration; heart failure; fluid overload
MeSH Terms: conditions — Heart Failure; Edema | interventions — Ultrafiltration

ARMS (2):
- Ultrafiltration (Experimental): Ultrafiltration treatment
  Interventions: Procedure: ultrafiltration
- Usual treatment (Active Comparator): Usual HF treatment
  Interventions: Procedure: ultrafiltration

INTERVENTIONS:
Procedure: ultrafiltration

SUMMARY:
Patients with severe congestive heart failure show increased fluid body content which is often resistant to conventional diuretic therapy. Therefore, chronic heart failure patients have frequent access to the emergency room and hospital for hemodynamic instability. Ultrafiltration is a simple renal replacement therapy which reduces fluid overload. The purpose of this study is to determine whether periodic ultrafiltration sessions maintain patients in stable clinical condition and reduce hospitalisations as well as access to emergency heart failure treatment.

DETAILED DESCRIPTION:
Patients with severe heart failure (New York Heart Association [NYHA] III-IV) and fluid overload will be randomized to ultrafiltration (UF group) or conventional medical treatment (Control group). Patients follow-up at least monthly visit for one year. Ultrafiltration will be repeated during follow-up in case of body weight gain due to fluid accumulation. Ultrafiltration will be performed during short term hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Severe heart failure (NYHA III-IV) with fluid overload
* Ejection fraction < 40%
* Estimated fluid overload > 4 kg

Exclusion Criteria:

* Severe renal insufficiency
* Acute pulmonary edema and/or cardiogenic shock

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
number of hospitalizations for heart failure | End of study

SECONDARY OUTCOMES:
long term major adverse clinical events including death | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, MD.PhD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

REFERENCES:
- [Derived] Marenzi G, Muratori M, Cosentino ER, Rinaldi ER, Donghi V, Milazzo V, Ferramosca E, Borghi C, Santoro A, Agostoni P. Continuous ultrafiltration for congestive heart failure: the CUORE trial. J Card Fail. 2014 Jan;20(1):9-17. doi: 10.1016/j.cardfail.2013.11.004. Epub 2013 Nov 20. PMID 24269855